CLINICAL TRIAL: NCT00806208
Title: Phase I Evaluation of Safety, Pharmacokinetics and Activity of Escalating Dose Levels of MEDI 507 in Patients Receiving Methylprednisolone for Initial Treatment of at Least Grade II Graft-Versus-Host Disease (GvHD)
Brief Title: Trial for Evaluation of Safety of Escalating Dose Levels of MEDI-507 in Patients for Treatment of at Least Grade II Graft-Versus-Host Disease (GvHD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: J. Bruce McClain, M.D., Medimmune Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP046
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-12

CONDITIONS: Graft-Versus-Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — siplizumab

ARMS (5):
- 1 (Active Comparator): MEDI 507 and Methylprednisolone
  Interventions: Drug: MEDI-507
- 2 (Active Comparator): MEDI-507 and Methylprednisolone
  Interventions: Drug: MEDI-507
- 3 (Active Comparator): MEDI-507 and Methylprednisolone
  Interventions: Drug: MEDI-507
- 4 (Active Comparator): MEDI-507 and Methylprednisolone
  Interventions: Drug: MEDI-507
- 5 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MEDI-507 — 0.012 mg/kg MEDI 507 and Methylprednisolone
  Arms: 1
Drug: MEDI-507 — 0.04 mg/kg MEDI 507 and Methylprednisolone
  Arms: 2
Drug: MEDI-507 — 0.12 mg/kg MEDI 507 and Methylprednisolone
  Arms: 3
Drug: MEDI-507 — 0.4 mg/kg MEDI 507 and Methylprednisolone
  Arms: 4
Other: Placebo — Placebo IV (alternative) study days 0, 3,6, and 9
  Arms: 5

SUMMARY:
A trial to assess safety of four doses of MEDI 507 combined with another drug for initial treatment of at least Grade II acute Graft-vs-Host Disease in recipients.

DETAILED DESCRIPTION:
The primary objective of this study is to assess safety of four dose levels of MEDI 507 combined with methylprednisolone for initial treatment of at least Grade II acute GvHD in stem cell or bone marrow allograft recipients.

ELIGIBILITY:
Inclusion Criteria:

1. allogeneic bone marrow or hematopoietic stem cell graft recipients
2. acute GvHD of at least Grade II severity
3. receipt of at least 2 mg/kg of methylprednisolone (or equivalent corticosteroid) within eight to 24 hours prior to initial receipt of study drug
4. evidence of engraftment (ANC over 1,000 cells/mm3)
5. histologic evidence of GvHD from biopsy performed during the current episode
6. receipt of GvHD prophylaxis of methotrexate, tacrolimus or cyclosporine
7. age at least 18 years
8. body weight under 130 kg
9. Both males and females are eligible, but females of childbearing potential, unless previously surgically sterilized, agree to use an effective method of birth control (e.g., abstinence, intrauterine contraceptive device, oral contraceptives, diaphragm or condom in combination with contraceptive jelly, cream or foam, Norplant7 or DepoProvera7) beginning with the first study injection and continuing through 60 days after the final study injection.

Exclusion Criteria:

1. previous receipt of MEDI 507
2. diagnosis of chronic GvHD
3. previous treatment with any anti-T-cell monoclonal antibodies such as OKT73 or daclizumab (Zenapax7)
4. receipt of antithymocyte globulin (ATGAM7 or other ATG) within 14 days
5. treatment with more than 0.3 mg/kg/day of methylprednisolone (or equivalent corticosteroid) for more than 72 hours for the treatment of GvHD
6. intolerance or history of intolerance to corticosteroids such that it is unlikely the patient will be able to complete at least ten days of corticosteroid therapy (2 mg/kg/day of methylprednisolone or equivalent)
7. more than one allogeneic bone marrow or hematopoietic stem cell allograft

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 1999-01; Primary Completion 2000-01 (Actual); Study Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
Safety; first infusion of study drug | Through Study Day 44

CONTACTS AND LOCATIONS:
Overall Officials: J. Bruce McClain, M.D., Study Director — MedImmune LLC
Locations (3):
- United States (3):
  - Washington University Medical Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Baylor Institute of Transplant Sciences, Dallas, Texas